CLINICAL TRIAL: NCT04315480
Title: Tocilizumab (RoActemra) as Early Treatment of Patients Affected by SARS-CoV2 (COVID-19) Infection With Severe Multifocal Interstitial Pneumonia
Brief Title: Tocilizumab for SARS-CoV2 (COVID-19) Severe Pneumonitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Azienda Ospedaliera Ospedali Riuniti Marche Nord (Unknown)
Responsible Party: Principal Investigator, Armando Gabrielli, Full Professor Internal Medicine, Università Politecnica delle Marche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOCICOV-1
Record Dates: First submitted 2020-03-14; First posted 2020-03-19 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: SARS Pneumonia
Keywords: Tocilizumab
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Simon's Two-stages Optimal Design
Masking Description: Radiologist will be blinded for sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — single intravenous administration 8mg/Kg

SUMMARY:
In a Phase 2 Simon's Optimal Two-Stages Design intravenous tocilizumab will be administered as single 8mg/Kg dose in patients affected by severe multifocal interstitial pneumonia correlated to SARS-CoV2 infection. Aim of the study is to test the hypothesis that an anti-IL6 treatment can be effective in calming the virus-induced cytokine storm, blocking deterioration of lung function or even promoting a rapid improvement of clinical conditions, preventing naso-tracheal intubation and/or death.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV2 Infection diagnosed by rt-PCR
* CT-scan confirmed multifocal interstitial pneumonia
* Need of oxygen therapy to maintain SO2>93%
* Worsening of lung involvement, defined as (one of the following criteria):

  * Worsening of oxygen saturation >3 percentage points or decrease in PaO2 >10%, with stable FiO2 in the last 24h
  * Need of increase FiO2 in order to maintain a stable SO2 or new onset need of mechanical ventilation in the last 24h
  * Increase in number and/or extension of pulmonary areas of consolidation

Exclusion Criteria:

* Age <18 ys and >90 ys
* Severe heart failure
* Bacterial Infection
* Haematological neoplasm
* Neutrophil count below 1000/mcl
* Platelet count below 50000/mcl
* ALT> x5UNL
* Inability to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-04-09 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
arrest in deterioration of pulmonary function | 7days
  rate of patients with no need in increase of FiO2 to maintain stable SO2 and no need of intubation
improving in pulmonary function | 7 days
  rate of patients with change of oxygen saturation >3 percentage points or >10% or decrease in FiO2 need or reduction in pulmonary consolidations >30% at HR CT-scan

SECONDARY OUTCOMES:
need of oro-tracheal intubation | +7 days
  rate of patients needed of intubation
death | 14days
  rate of patients dead

CONTACTS AND LOCATIONS:
Locations (1):
- Università Politecnica delle Marche, Ancona, AN, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian S, Hu W, Niu L, Liu H, Xu H, Xiao SY. Pulmonary Pathology of Early-Phase 2019 Novel Coronavirus (COVID-19) Pneumonia in Two Patients With Lung Cancer. J Thorac Oncol. 2020 May;15(5):700-704. doi: 10.1016/j.jtho.2020.02.010. Epub 2020 Feb 28. PMID 32114094
- [Background] Ashour HM, Elkhatib WF, Rahman MM, Elshabrawy HA. Insights into the Recent 2019 Novel Coronavirus (SARS-CoV-2) in Light of Past Human Coronavirus Outbreaks. Pathogens. 2020 Mar 4;9(3):186. doi: 10.3390/pathogens9030186. PMID 32143502
- [Background] Channappanavar R, Perlman S. Pathogenic human coronavirus infections: causes and consequences of cytokine storm and immunopathology. Semin Immunopathol. 2017 Jul;39(5):529-539. doi: 10.1007/s00281-017-0629-x. Epub 2017 May 2. PMID 28466096
- [Background] Zumla A, Ippolito G, Ntoumi F, Seyfert-Margolies V, Nagu TJ, Cirillo D, Chakaya JM, Marais B, Maeurer M. Host-directed therapies and holistic care for tuberculosis. Lancet Respir Med. 2020 Apr;8(4):337-340. doi: 10.1016/S2213-2600(20)30078-3. Epub 2020 Feb 27. No abstract available. PMID 32113574
- [Derived] Sabbatinelli J, Giuliani A, Matacchione G, Latini S, Laprovitera N, Pomponio G, Ferrarini A, Svegliati Baroni S, Pavani M, Moretti M, Gabrielli A, Procopio AD, Ferracin M, Bonafe M, Olivieri F. Decreased serum levels of the inflammaging marker miR-146a are associated with clinical non-response to tocilizumab in COVID-19 patients. Mech Ageing Dev. 2021 Jan;193:111413. doi: 10.1016/j.mad.2020.111413. Epub 2020 Dec 8. PMID 33307107

DOCUMENTS (1):
  • Study Protocol (2020-03-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT04315480/Prot_000.pdf